CLINICAL TRIAL: NCT07132944
Title: Development and Feasibility of a Function-focused Transitional Care Intervention to Support Functional Recovery in Older Veterans
Brief Title: Development and Feasibility of CTraC-FIT
Acronym: CTraC-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RRD9-002-24W; 1IK2RD000454-01A1 (Other Grant/Funding Number: Rehabilitation Research and Development)
Record Dates: First submitted 2025-07-29; First posted 2025-08-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Functional Impairment; Functional Performance
Keywords: Physical function; Transitional care; Function-focused care; Function; Care Transition; Physical performance; Functional performance; Health care transition; Transition of care

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a pilot randomized controlled trial (RCT) to evaluate the feasibility, acceptability, and preliminary effects of the CTraC-FIT protocol. Participants will be randomized into two groups: CTraC-FIT intervention and control group receiving enhanced usual care (EUC).
Who Masked: Participant
Masking Description: Given the nature of the intervention, it is not feasible to use double blinding where both participants and assessors are unaware of group assignments. Instead, a single-blind design will be employed where the participants are not aware of their specific group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTraC-FIT (Experimental): The intervention arm involves participants receiving a structured transitional care intervention (CTraC-FIT) administered by a trained nurse case manager via phone or VA Video Connect, aimed at improving functional abilities and reducing hospital readmissions.
  Interventions: Other: CTraC-FIT
- Enhanced Usual Care (Other): The Enhanced Usual Care (EUC) arm involves participants receiving the standard care provided by their assigned Veterans Affairs Boston Healthcare System (VABHS) inpatient and outpatient teams.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: CTraC-FIT — The intervention is designed to support Veterans at high risk of readmission with comprehensive transitional care that includes:
  Structured Follow-Ups: Regularly scheduled follow-up calls to monitor the patient's progress, address any issues, and provide ongoing support.
  Health Coaching: Personalized coaching to help Veterans manage their health conditions, adhere to treatment plans, and make lifestyle changes that can improve their overall health.
  Care Coordination: Assistance with navigating the healthcare system, facilitating appointments, and ensuring that the Veteran receives all necessary post-discharge services.
  The intervention arm aims to improve functional abilities and reduce hospital readmissions by providing tailored support based on the unique needs of each participant. The CTraC NCM will follow a standardized protocol to ensure consistent and effective delivery of the intervention across all participants in this group.
  Other Names: Coordinated Transitional Care
  Arms: CTraC-FIT
Other: Enhanced Usual Care — The Enhanced Usual Care (EUC) arm involves participants receiving the standard care provided by their assigned Veterans Affairs Boston Healthcare System (VABHS) inpatient and outpatient teams. This includes routine medical evaluations, treatments, and follow-up appointments as typically recommended by their healthcare providers. In addition to receiving standard care, participants in the EUC group will undergo baseline, endpoint, and 3-month follow-up assessments as part of the study protocol.
  For participants with intermediate functional ability (SPPB score of 7-9), no additional intervention will be provided after randomization to the control group. However, for participants with low functional ability (SPPB score of 0-6), a safety protocol will be activated to notify their assigned inpatient medical team (e.g., hospitalist, social worker) about the participant's risk of functional decline, ensuring that appropriate support and referrals are provided if needed.
  Other Names: EUC
  Arms: Enhanced Usual Care

SUMMARY:
Functional decline after hospitalization is a serious concern for older Veterans, often leading to loss of independence and disability. VA's nurse-led Coordinated Transitional Care (CTraC) program has demonstrated success in improving care transitions, but currently lacks targeted assessment and intervention to support Veterans' functional recovery. This project aims to develop and test a function-focused CTraC protocol (CTraC-FIT) to address this critical gap and optimize functional outcomes for Veterans transitioning from hospital to home. By integrating evidence-based functional assessment and intervention strategies into the CTraC protocol, this project aims to empower Veterans to regain and maintain their independence and improve their quality of life.

DETAILED DESCRIPTION:
Nearly two-thirds of older adults experience significant functional decline after hospital discharge, resulting in loss of independence, institutionalization, and even death. Functional decline (i.e., loss of physical or cognitive ability that makes it difficult or impossible to perform activities of daily living) often occurs after hospital discharge due to a complex interplay between pre-existing health conditions, physiological stressors, and reduced mobility and activity levels during hospitalization. Veterans are at particular risk of functional decline as they experience a disproportionate burden of physical and psychological conditions compared to their non-Veteran peers. Transitions from hospital to home serve as critical junctures to address Veterans' functional needs, but many patients are discharged without a comprehensive functional evaluation. Even when evaluation occurs, discharge plans often fail to translate into effective care delivery, creating a concerning gap between planned and actual support after hospitalization.

The Coordinated Transitional Care (CTraC) program is a potential foundation on which to build a protocol that meets Veterans' rehabilitative care needs during and after discharge. CTraC is a nurse-led transitional care program developed to improve Veterans' transitions to the community after hospitalization. CTraC aims to address key components of transitional care: (1) care planning and communication; (2) medical follow-up; (3) education on symptom management; and (4) medication safety/management. In this model, the CTraC nurse identifies and meets Veterans at high risk of readmission, helps optimize their discharge planning, and then delivers a protocolized phone-based intervention for up to 30 days. CTraC has demonstrated significant benefits to VA, including a 50% reduction in readmissions, resolution of medication discrepancies for more than half of enrolled patients, and cost savings. Yet, the existing CTraC protocol misses a critical opportunity to include functional assessment and intervention to support Veterans' functional recovery.

The goal of this CDA-2 proposal is to develop and test a function-focused protocol for VA's CTraC program. The aim is to leverage CTraC's established success and infrastructure to comprehensively address Veterans' rehabilitation needs after hospitalization and optimize their functional recovery and independence during the transition from hospital to home. Specifically, this project aims to:

Aim 1: Develop & refine CTraC-FIT (Functional Independence aT home) for Veterans at risk of functional decline transitioning from hospital to home. (1a) Develop CTraC-FIT to support Veterans' functional recovery based on input from clinicians (n=15) across hospital and outpatient settings (e.g., CTraC NCMs, inpatient providers, primary care providers, physical therapists, and occupational therapists). (1b) Conduct a nonrandomized, preliminary pilot of the CTraC-FIT intervention (n=5 Veterans) and collect qualitative feedback from Veterans and the CTraC NCM to refine the intervention protocol and study procedures, as well as address any unanticipated barriers before pilot testing.

Aim 2: Examine the feasibility and acceptability of CTraC-FIT in a pilot randomized controlled trial via randomization of n=40 Veterans to either CTraC-FIT (n=20) or an enhanced usual care condition (n=20). The primary outcomes will be feasibility and acceptability of the intervention protocol and study procedures. Feasibility and acceptability of the intervention protocol will be measured via survey and qualitative interviews with Veterans, and surveys with clinicians (n~20). Feasibility of the study procedures will be assessed via data logs (e.g., recruitment, enrollment, retention, adherence, randomization, and fidelity). Secondary outcomes will include Veterans' self-reported quality of life, social and cognitive function as well as self-reported and performance-based physical function measured at baseline, post-intervention, and 3-months post-intervention.]

ELIGIBILITY:
Inclusion Criteria:

* .Age > or = 65 years
* Score of > 3 on Vulnerable Elders Survey, (VES-13)
* Score of 4-9 on Short Physical Performance Battery (SPPB)
* Able to provide informed consent

Exclusion Criteria:

* Admitted to VA Boston for acute psychiatric are or substance abuse detoxification
* Plan to discharge anywhere except home (e.g., assisted living, group home, or skilled nursing facility)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | Endpoint (Day 30)
  We will measure Veteran satisfaction using the Client Satisfaction Questionnaire (CSQ-8), a validated tool that assesses satisfaction with various aspects of service delivery, including the quality of care, helpfulness of staff, and overall experience.
Perceived Characteristics of Intervention Scale | Endpoint (Day 30)
  We will use the Perceived Characteristics of Intervention Scale (PCIS) to understand clinicians' perspectives on the acceptability of the CTraC-FIT intervention. The PCIS is a validated tool designed to assess key factors influencing the acceptability of an intervention from the perspective of healthcare providers. Developed within VA, the scale assesses the overall acceptability of the intervention by examining whether it is perceived as beneficial, feasible, and compatible with existing practices.
Enrollment | Baseline (Day 1)
  Assessed by the proportion of those screened who enroll in the study, as well as the number of participants enrolled each month. This data will be sourced from the project database.
Recruitment | Baseline (Day 1)
  Measured by the proportion of participants approached who agree to screening. This data will be sourced from the project database.
Retention | Endpoint (Day 30); 3-Month
  Proportion of enrolled participants who complete the endpoint assessment and the 3-month follow-up. This data will be sourced from the project database.
Adherence | Endpoint (Day 30); 3 Month
  We will use a combination of metrics to determine adherence, including:
  The proportion of completed phone or VVC (Video Visit Communication) calls The proportion of participants who establish functional goals The proportion of participants who achieve at least 50% of their goals The proportion of participants with a documented functional recovery care plan within 72 hours post-discharge This data will be sourced from the project database.
Fidelity | Endpoint (Day 30)
  Assessed by compliance with the CTraC-FIT fidelity checklist. This data will be sourced from the project database.

SECONDARY OUTCOMES:
Performance-based Physical Function | Baseline (Day 1), Endpoint (Day 30), 3 Month
  We will use the Short Physical Performance Battery (SPPB) to measure performance-based physical function over time. The SPPB's strong psychometric properties and ability to predict future disability and adverse events make it a valuable tool for evaluating the impact of the CTraC-FIT intervention on physical function and mobility.
Self-reported Physical, Cognitive, and Social Function | Baseline (Day 1), Endpoint (Day 30), 3 Month
  We will use the World Health Organization Disability Assessment Schedule (WHODAS) 2.0 to measure physical, cognitive, and social function over the past 30 days, offering a comprehensive evaluation of function and disability. This self-report tool uses a 5-point Likert scale to assess difficulties in six domains: understanding and cognition, mobility, self-care, getting along, life activities, and participation.
Quality of Life | Baseline (Day 1), Endpoint (Day 30), 3 Month
  We will use the World Health Organization Quality of Life-BREF (WHOQOL-BREF) self-report instrument to assess and produce scores representative of quality of life in the domains of physical health, psychological health, social relationships, and environment in a 2-week timeframe. The WHOQOL-BREF's strong psychometric properties and comprehensive coverage of quality-of-life domains make it a valuable tool for understanding the potential impact of the CTraC-FIT intervention.

OTHER OUTCOMES:
Functional Ability Screener | Pre-baseline - during CTraC program enrollment
  We will use a self-reported measure of risk of functional decline-the Vulnerable Elders Survey and a performance-based measure of physical functional impairment-the Short Physical Performance Battery (SPPB). Veterans eligible for study participation will have both a score of ≥ 3 on the VES-13 indicating an increased risk of functional decline and a score of 4-9 on the SPPB.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Madrigal, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No